CLINICAL TRIAL: NCT04079621
Title: Short Course Radical Cure of P.Vivax in Nepal- a Randomized Controlled Trial
Brief Title: Short Course Radical Cure of P. Vivax Malaria in Nepal
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Collaborators: Tribhuvan University, Nepal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIRIN
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Malaria; Malaria, Vivax; Malaria,Falciparum
MeSH Terms: conditions — Malaria; Malaria, Vivax; Malaria, Falciparum | interventions — Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- (P.f) (Experimental): patients with falciparum malaria will receive artemether-lumefantrine (AL) twice daily over three days plus a low dose course of primaquine (PQ) (3.5mg/kg total dose) given 7 days during schizontocidal treatment
  Interventions: Drug: primaquine
- (P.v) (Experimental): patients with vivax malaria will receive chloroquine (CQ) daily for three days plus a low dose course of PQ (3.5mg/kg total dose) given over 7 days during schizontocidal treatment.
  Interventions: Drug: primaquine
- Standard care (P.f) (No Intervention): patients with falciparum malaria will receive artemether-lumefantrine (AL) twice daily over three days (plus a single dose PQ)
- Standard care (P.v) (No Intervention): patients with vivax malaria will receive chloroquine (CQ) daily for three days plus a low dose course of PQ (total dose 3.5mg/kg) over 14 days

INTERVENTIONS:
Drug: primaquine — Primaquine regimen over 7 days (0.5mg/kg/day for 7 days)
  Other Names: Jasoprim, Malirid, Neo-Quipenyl, Pimaquin, Pmq, Primachina, Primacin, Primaquina, Primaquine, Primaquine diphosphate, Primaquine Phosphate, and Remaquin
  Arms: (P.f); (P.v)

SUMMARY:
This study is designed as a multicentre randomized, open label trial to assess the safety and efficacy of a low dose short course PQ treatment (3.5mg/kg total dose given over 7 days) in glucose-6-phosphate dehydrogenase (G6PD) normal patients with P.vivax and P falciparum to reduce the risk of subsequent P.vivax episodes.

DETAILED DESCRIPTION:
Plasmodium vivax is associated with recurrent infections weeks or months following the acute infection due to reactivation of dormant liver stages. Recurrent infections can be associated with a febrile illness, cumulative risk of severe anaemia, direct and indirect mortality, and are the most important source of onward transmission of the parasite.

In co-endemic areas, there is a very high risk (up to 50%) of patients representing with P.vivax malaria following treatment of P falciparum. Hence, in co-endemic regions there is a strong rationale for eradicating P.vivax hypnozoites from the liver in patients presenting with uncomplicated P. falciparum infections.

The recently completed multicentre IMPROV study compared the efficacy of a 7 day PQ regimen (1.0mg/kg/day for 7 days) with a 14 day regimen (0.5mg/kg/day for 14 days). The 7 day PQ regimen was non-inferior to the 14 day regimen and 5 times more efficacious at reducing P.vivax recurrence than the control.

This study is designed as a multicentre randomized, open label trial to assess the safety and efficacy of a low dose short course PQ treatment (3.5mg/kg total dose given over 7 days) in G6PD normal patients with P.vivax and P falciparum to reduce the risk of subsequent P.vivax episodes.

ELIGIBILITY:
Inclusion Criteria:

* P. falciparum and/or vivax infection
* Fever (axillary temperature ≥37.5⁰C) or history of fever in preceding 48 hours
* Age >1 years
* G6PD normal by Rapid Diagnostic Test (RDT) as per national guidelines
* Written informed consent
* Able to comply with all study procedures and timelines

Exclusion Criteria:

* General danger signs or symptoms of severe malaria
* Anaemia, defined as Hb <8g/dl
* Pregnant women as determined by Urine β-HCG pregnancy test
* Breast feeding women
* Known hypersensitivity to any of the drugs given
* Regular use of drugs with haemolytic potential
* Blood transfusion within the last 4 months

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence Risk of P. vivax relapse at month 6 | 6 months
  The incidence risk of symptomatic P. vivax malaria at month 6 in patients enrolled with P. vivax and P. falciparum infection.

SECONDARY OUTCOMES:
The incidence risk of symptomatic P. vivax malaria at month 6 in patients enrolled with P. vivax | 6 months
The incidence risk of symptomatic P. vivax malaria at month 6 in patients enrolled with P. falciparum | 6 month
The incidence risk of symptomatic P. vivax malaria at day 28 in patients enrolled with P. falciparum and vivax malaria infection | Day 28
The incidence risk of all (symptomatic and asymptomatic) P. vivax malaria at day 28 in patients enrolled with P. falciparum and vivax malaria infection | Day 28
The incidence risk of asymptomatic P. vivax malaria at day 28 in patients enrolled with P. falciparum and vivax malaria infection | Day 28

OTHER OUTCOMES:
The proportion of patients vomiting their medication within 1 hour of administration | 1 h
The proportion of patients vomiting any of their PQ doses during the supervised course | 7 - 14days
The proportion of adverse events and serious adverse events | 6 month
The incidence risk of severe anaemia (Hb<7g/dl) and/or the risk for blood transfusion | 6 month
Risk of greater than 25% fall in haemoglobin on any day of treatment | 7-14days
The incidence risk of an acute drop in Hb of >5g/dl during PQ treatment | 7-14days

CONTACTS AND LOCATIONS:
Overall Officials: Kamala Ley-Thriemer, MD, PhD, Principal Investigator — Menzies School of Health Research
Locations (2):
- Nepal (2):
  - Malakheti Hospital, Malakheti
  - Tikapur Hospital, Ṭikāpur

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and Statistical Analysis Plan will be made available to others. Data collected for the study, including individual patient data and the final trial dataset are reserved for the chief investigator and co-investigators of the trial. The trial will be reported in accordance with the Consolidated Standards of Reporting Trials (CONSORT) guidelines. Trial results will be published in peer-reviewed open access journals and disseminated to trial stakeholders, including participants, as per ethical guidelines.
Supporting Information: Study Protocol, SAP
Access Criteria: The data are available for access via the WorldWide Antimalarial Resistance Network (WWARN.org). Requests for access will be reviewed by a Data Access Committee to ensure that use of data protects the interests of the participants and researchers according to the terms of ethics approval and principles of equitable data sharing. Requests can be submitted by email to malariaDAC@iddo.org via the Data Access Form available at WWARN.org/accessing-data. The WWARN is registered with the Registry of Research Data Repositories (re3data.org).
URL: http://WWARN.org/accessing-data